CLINICAL TRIAL: NCT04100187
Title: Phase I Study of T Cells Expressing an Anti-CD19 Chimeric Receptor in Children and Young Adults With B Cell Leukemia
Brief Title: Immunotherapy With CD19 CAR T-cells for B-Cell Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kecellitics Biotech Company Ltd (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kece-1
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Leukemia
Keywords: CAR-T; Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental:3 (Experimental): Leukemia treated with chimeric antigen receptor modified T cells(Anti-CD19-CAR) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR

INTERVENTIONS:
Biological: Anti-CD19-CAR — Cells extracted, followed by induction chemotherapy before CD19-CAR infusion (dose escalation.)

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of CD19 Chimeric Antigen Receptor (CAR) redirected autologous T-cells in patients with high risk, relapsed CD19+ haematological malignancies.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19 Chimeric Antigen Receptor (CAR) T-cells (CD19 CAR T-cells) in patients with high risk, relapsed CD19+ Leukemia. Following informed consent and registration to the trial, patients will undergo an unstimulated leukapheresis for the generation of the CD19 CAR Tcells.

Patients will receive the CD19CAR T-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CAR T-cells in patients with high risk relapsed CD19+ Leukemia

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell Leukemia.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 2 years to 70 years.
5. CD19 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 30% by flow cytometry.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.
12. Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to trial

Exclusion Criteria:

1. KPS<50.
2. Patients are allergic to cytokines.
3. Uncontrolled active infection.
4. Acute or chronic GVHD.
5. Treated with T cell inhibitor.
6. Pregnancy and nursing females.
7. HIV/HBV/HCV Infection.
8. Other situations we think improper for the research.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of each patient | 3 years
  Determine the toxicity profile of the CD19 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.
Survival time of Anti-CD19 CAR T cells in vivo | 3 years
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Antitumor Effects | Every 3 months post treatment up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.
Maximum tolerated dose (MTD) of CD19 targeted CAR T cells. | 4 weeks
  Maximum tolerated dose (MTD) of CD19 targeted CAR T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Li xiangqun, Study Chair — Kecellitics Biotech Company Ltd